CLINICAL TRIAL: NCT02943421
Title: Evaluation of the Efficacy of Transverse B-Lynch in Management of Placenta Accreta
Brief Title: Transverse B-Lynch in Management of Placenta Accreta
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Other Study IDs: MAP
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Decrease Maternal Morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Transverse B-Lynch suture

SUMMARY:
Placenta accreta is considered a severe pregnancy complication that may be associated with massive and potentially life-threatening intrapartum and postpartum hemorrhage. Life-threatening bleeding is the most common complication to be associated with this condition; the average blood loss at time of delivery is reported to be 3000-5500 mL, which leads to significant postoperative morbidity and death.

ELIGIBILITY:
Inclusion Criteria:

1. All pregnant women with placenta previa as diagnosed by ultrasound with suspicion of abnormal placentation by Doppler us, confirmed intraoperatively undergoing either emergent or elective cesarean

Exclusion Criteria:

1. Patients who will be managed by hysterectomy
2. Patients who will be managed by conservative leaving the placenta in-situ

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the study encompassing women managed by conservative transverse B-Lynch during cesarean section due to placenta accreta
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-02-03 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Estimated intraoperative blood loss | 30 min

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No